CLINICAL TRIAL: NCT00551057
Title: Expression of Inflammatory Proteins in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Dr. Marc Schiesser, University Hospital Zurich/VIS Klinik f. Viszeralchirurgie
Other Study IDs: 13-2007
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2007-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — To investigate the expression of different inflammatory proteins in cancer and normal pancreatic tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Expression type — to investigate the expression of different inflammatory proteins in cancer and normal pancreatic tissue

SUMMARY:
The purpose of this trial is to investigate the expression of different inflammatory proteins in cancer and normal pancreatic tissue.

DETAILED DESCRIPTION:
Purpose: to investigate the expression of different inflammatory proteins in cancer and normal pancreatic tissue

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* Patients with pancreatic cancer or chronic pancreatitis

Exclusion criteria:

* Patients with alpha 1-antitrypsin deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer or chronic pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schiesser, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich Department of Surgery, Zurich, Switzerland